CLINICAL TRIAL: NCT01932970
Title: A Multicenter, Multiple-dose, Single-arm Study to Switch Hemodialysis Subjects With Secondary Hyperparathyroidism From Oral Cinacalcet HCl to Intravenous AMG 416
Brief Title: Study to Assess the Impact on Calcium Levels When Hemodialysis Patients With Secondary Hyperparathyroidism (SHPT) Switch From Cinacalcet to Etelcalcetide
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20120359; 2013-000964-28 (EudraCT Number); KAI-4169 (Other: KAI Pharmaceuticals (wholly owned subsidiary of Amgen Inc.))
Record Dates: First submitted 2013-08-28; First posted 2013-08-30 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-09

CONDITIONS: Hyperparathyroidism, Secondary
Keywords: Secondary Hyperparathyroidism (SHPT), chronic kidney disease (CKD), hemodialysis, parathyroid hormone (PTH), hypocalcemia, bone and mineral metabolism
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Renal Insufficiency, Chronic; Hypocalcemia | interventions — etelcalcetide hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Etelcalcetide (Experimental): Participants were treated with 5 mg etelcalcetide administered by intravenous bolus injection at the end of each hemodialysis session three times per week (TIW) for 4 weeks.
  Interventions: Drug: Etelcalcetide

INTERVENTIONS:
Drug: Etelcalcetide — Etelcalcetide is provided as a sterile lyophilized powder to be reconstituted with sterile water for injection.
  Other Names: KAI 4169; AMG 416; Parsabiv™

SUMMARY:
This is a multicenter, multiple-dose, single-arm, open-label study to assess the impact on serum corrected calcium levels when switching patients from cinacalcet to etelcalcetide (AMG 416).

ELIGIBILITY:
Inclusion Criteria

* Subject is 18 years of age or older at the time of informed consent.
* Subject must be receiving maintenance hemodialysis 3 times weekly for at least 8 weeks.
* Subject must have SHPT as defined by having a mean of 3 consecutive central laboratory screening predialysis serum parathyroid hormone (PTH) values ≥ 200 pg/mL, with measurements obtained from 3 different calendar weeks in the 4-week screening period while receiving cinacalcet.
* Subject must have a mean of 3 consecutive central laboratory screening predialysis serum corrected calcium (cCa) values ≥ 7.5 mg/dL, with measurements obtained from 3 different calendar weeks in the 4-week screening period while receiving cinacalcet.
* Subject must be on a stable dose of cinacalcet before screening (defined as no dose change within the 4 weeks prior to screening).
* Other Inclusion Criteria may apply.

Exclusion Criteria

* Currently receiving treatment in another investigational device or drug study, or less than 30 days since ending treatment on another investigational device or drug study(s).
* Subject has received AMG 416 in a prior clinical trial of AMG 416 (also known as KAI-4169).
* Subject has known sensitivity to any of the products or components of AMG 416 to be administered during dosing.
* Subject is unwilling to use effective contraception during the study, and for women, up to a period of up to 3 months after the last dose of AMG 416.
* Subject is pregnant or nursing.
* Anticipated or scheduled parathyroidectomy during the study period.
* Subject has received a parathyroidectomy within 6 months prior to dosing.
* Other Exclusion Criteria may apply.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2013-08-12 (Actual); Primary Completion 2014-01-14 (Actual); Study Completion 2017-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (40):
- United States (40):
  - Research Site, Alhambra, California
  - Research Site, Azusa, California
  - Research Site, Bakersfield, California
  - Research Site, Chula Vista, California
  - Research Site, La Mesa, California
  - Research Site, Los Angeles, California
  - Research Site, Lynwood, California
  - Research Site, Riverside, California
  - Research Site, Whittier, California
  - Research Site, Arvada, Colorado
  - Research Site, North Haven, Connecticut
  - Research Site, Coral Springs, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Miami, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Pinecrest, Florida
  - Research Site, Tampa, Florida
  - Research Site, Augusta, Georgia
  - Research Site, Evergreen Park, Illinois
  - Research Site, Michigan City, Indiana
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Lafayette, Louisiana
  - Research Site, Columbus, Mississippi
  - Research Site, Gulfport, Mississippi
  - Research Site, Farmington, Missouri
  - Research Site, Kansas City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Portsmouth, New Hampshire
  - Research Site, Eatontown, New Jersey
  - Research Site, College Point, New York
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Orangeburg, South Carolina
  - Research Site, Arlington, Texas
  - Research Site, Greenville, Texas
  - Research Site, Houston, Texas
  - Research Site, McAllen, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Fairfax, Virginia
  - Research Site, Hampton, Virginia

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 33 centers in the United States. Participants were enrolled from 1 September 2013 to 9 December 2013.
  Participants were required to be on a stable dose of daily oral cinacalcet for a minimum of 4 weeks before screening, and during the 4 weeks of screening.
Pre-assignment Details: Upon enrollment, participants underwent a washout period of a minimum of 7 days, wherein no cinacalcet use was allowed. Participants who had a serum corrected calcium ≥ 8.3 mg/dL during the washout period entered the treatment phase and were categorized based on their pre-washout, screening cinacalcet daily dose level (30 mg, 60 mg or ≥ 90 mg).
Period: Overall Study
Arm/Group | Etelcalcetide
Started | 158 (Includes all participants who enrolled into the washout period.)
Received Treatment | 148 (Includes participants who completed the washout period and received etelcalcetide)
Completed | 140
Not Completed | 18
Not completed — Withdrawal by Subject | 5
Not completed — Death | 1
Not completed — Lost to Follow-up | 2
Not completed — Protocol Specified Criteria | 10

BASELINE CHARACTERISTICS:
Population: Full analysis set includes iall participants who enrolled into the study and had at least one dose of etelcalcetide and at least one post-baseline serum corrected calcium value.
Arm/Group | Etelcalcetide
Number analyzed (Participants) | 147
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (14.0)
Age, Customized [Number; unit: participants]
  < 65 years | 106
  ≥ 65 years | 41
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 92
Race [Number; unit: participants]
  American Indian or Alaska Native | 1
  Asian | 12
  Black (or African American) | 68
  Native Hawaiian or Other Pacific Islander | 2
  White | 64
Ethnicity [Number; unit: participants]
  Hispanic/Latino | 39
  Not Hispanic/Latino | 108
Corrected Calcium [Mean (Standard Deviation); unit: mg/dL] — When albumin was less than 4.0 g/dL, the calcium level was corrected according to the following formula:
  Corrected calcium (cCa) (mg/dL) = total Ca (mg/dL) + (4 - albumin [g/dL]) * 0.8.
  mg/dL | 9.81 (0.75)
Parathyroid Hormone [Mean (Standard Deviation); unit: pg/mL] — Data available for 140 participants
  pg/mL | 786.3 (467.8)
Phosphorus [Mean (Standard Deviation); unit: mg/dL] — Data available for 135 participants
  mg/dL | 5.88 (1.71)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Serum Corrected Calcium < 7.5 mg/dL During the 4-week Treatment Period
Time Frame: 4 weeks
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etelcalcetide
Number analyzed (Participants) | 147
percentage of participants | 0.7 [0.0 to 3.7]

2. Secondary Outcome: Percent Change From Baseline in Parathyroid Hormone During the Treatment Period
Time Frame: Baseline and weeks 2, 3 and 4
Population: Full analysis set with available data at each time point
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Etelcalcetide
Number analyzed (Participants) | 140
percent change
  Week 2 (n = 125) | -3.9 (2.6)
  Week 3 (n = 131) | -7.8 (3.1)
  Week 4 (n = 123) | -10.9 (2.9)

3. Secondary Outcome: Percentage of Participants With Serum Corrected Calcium < 8.3 mg/dL During the 4-week Treatment Period
Time Frame: 4 weeks
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etelcalcetide
Number analyzed (Participants) | 147
percentage of participants | 15.6 [10.2 to 22.5]

4. Other Pre Specified Outcome: Number of Participants With Adverse Events
Time Frame: From the first dose of study drug up to 30 days after the last dose; 8 weeks
Population: All participants who received at least one dose of study drug
Measure: Number; unit: participants
Arm/Group | Etelcalcetide
Number analyzed (Participants) | 148
participants
  Any adverse event (AE) | 72
  Serious adverse event (SAE) | 17
  AE leading to discontinuation of etelcalcetide | 2
  Fatal adverse event | 1
  Treatment-related adverse event | 11

5. Other Pre Specified Outcome: Percentage of Participants With Symptomatic Hypocalcemia During the 4-week Treatment Period
Description: Hpocalcemia was used for events of decreased calcium accompanied by clinical signs and symptoms of hypocalcemia.
Time Frame: From the first dose of study drug up to 30 days after the last dose; 8 weeks
Population: Participants who received at least one dose of study drug
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etelcalcetide
Number analyzed (Participants) | 148
percentage of participants | 0.0 [0.0 to 2.5]

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to 30 days after the last dose; up to 8 weeks
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Etelcalcetide
Serious Adverse Events (participants affected / at risk) | 17/148
Other Adverse Events (participants affected / at risk) | 0/148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etelcalcetide (N=148)
Acute myocardial infarction (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Asthenia (General disorders) | 1
Chest pain (General disorders) | 1
Bile duct obstruction (Hepatobiliary disorders) | 1
Arteriovenous graft site infection (Infections and infestations) | 1
Biliary sepsis (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Staphylococcal bacteraemia (Infections and infestations) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Procedural hypotension (Injury, poisoning and procedural complications) | 1
Blood glucose increased (Investigations) | 1
Fluid overload (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.